CLINICAL TRIAL: NCT01376609
Title: A MRI-based Study of Ischaemic Penumbra: the Correlation Between Outcome and Infarct Growth in Patients With Acute Ischemic Stroke
Brief Title: The Correlation Between Outcome and Infarct Growth in Patients With Acute Ischemic Stroke
Acronym: COIG
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Hospital of Traditional Chinese Medicine (Other)
Collaborators: Beijing University of Chinese Medicine (Other)
Responsible Party: Jianghai Ruan, Dept.of Neurology，Beijing Dongfang Hospital, Beijing University of Chinese Traditional Medicine,Beijing,China
Other Study IDs: BUCM-002H-ND
Record Dates: First submitted 2011-06-17; First posted 2011-06-20 (Estimated); Last update posted 2011-08-01 (Estimated); Status verified 2011-06

CONDITIONS: Ischemic Stroke
Keywords: Stroke; Ischaemic Stroke; Cerebral Infarction; Cerebrovascular Disorders; Brain Diseases; Nervous System Diseases; Vascular Diseases; Brain Infarction; Brain Ischemia; mismatch; PWI/DWI mismatch; ischaemic penumbra; image analysis
MeSH Terms: conditions — Ischemic Stroke; Stroke; Cerebral Infarction; Cerebrovascular Disorders; Brain Diseases; Nervous System Diseases; Vascular Diseases; Brain Infarction; Brain Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Previous research has shown there wasn't inevitable relationship between mismatch area and infarct growth according to Volumetric-subtraction mismatch volume.The recently published on Stroke paper has proposed Coregistration mismatch to calculate the mismatch to replace ischaemic penumbra, and it reignites hope for clinical application of the PWI/DWI mismatch. But the correlation between the mismatch, calculated by Coregistration mismatch method,and the clinical outcome of the patients with acute ischemic stroke is still unknown. so the investigators plan to conduct a prospective observational cohort study.

DETAILED DESCRIPTION:
NIHSS,mRS and MR PWI/DWI/MRA are performed within 48 hours of stroke onset and final MR T2/flair image at ≈1 month. And then,Volumetric-subtraction mismatch and Coregistered mismatch will be calculated,respectively.finally,we will assess and compare the Volumetric-subtraction mismatch and Coregistered mismatch, and to clarify which method match the clinical outcome more better.

ELIGIBILITY:
Inclusion Criteria:

* Aged eighteen or above
* Acute middle cerebral artery ischemic stroke
* Stroke onset within 48 hours
* Included a complete set of initial MR images and final outcome MR images up to 1 months

Exclusion Criteria:

* History of stroke in the past 6 weeks
* Pre-existing neurological or psychiatric disease that could confound the study results such as a pre-stroke mRS score greater than 3
* CT evidence of the following conditions before enrollment:

Significant mass effect with midline shift Evidence of intracranial hemorrhage

* With contraindication to MR such as severe allergy to contrast media

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischaemic stroke admitted to ASU.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-03 (Estimated); Study Completion 2013-08 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Jianghai Ruan, Beijing, Beijing Municipality, China